CLINICAL TRIAL: NCT04230551
Title: Reverse Remodeling After PTSMA in Severe But ASympTomAtic LVOT Obstruction (RASTA Study)
Brief Title: Reverse Remodeling After PTSMA in Severe But Asymptomatic LVOT Obstruction
Acronym: RASTA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, J.M. ten Berg, Principal Investigator, St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RASTA_V6
Record Dates: First submitted 2019-12-31; First posted 2020-01-18 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: HOCM, Hypertrophic Obstructive Cardiomyopathy; LVOTO - Left Ventricular Outflow Tract Obstruction; Remodeling, Ventricular
Keywords: HOCM; Hypertrophic Obstructive Cardiomyopathy; Left Ventricular Outflow Tract Obstruction; Adverse Remodeling; Reverse Remodeling; Alcohol Septal Ablation; Percutaneous Transluminal Septal Myocardial Ablation; PTSMA; Extracellular Volume Fraction; Global Longitudinal Strain; Deformation Imaging; 4D Velocity Mapping
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Ventricular Outflow Obstruction, Left; Ventricular Remodeling | interventions — Ethanol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Technicians and/or imaging cardiologists involved in image analysis will not be informed about the procedure in order to have an unbiased analysis at baseline. At follow-up, treated patients will have akinetic/infarcted proximal septum that will be noticed during image acquisition. However, the pre-PTSMA status (symptomatic vs. asymptomatic) will be blinded for the analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reference Group (Active Comparator): Five symptomatic HOCM patients with severe LVOT obstruction will undergo PTSMA
  Interventions: Procedure: PTSMA
- Study Group (Experimental): Five asymptomatic HOCM patients with severe LVOT obstruction will undergo PTSMA
  Interventions: Procedure: PTSMA
- Observation Group (No Intervention): Five asymptomatic HOCM patients with severe LVOT obstruction will not undergo PTSMA

INTERVENTIONS:
Procedure: PTSMA — Alcohol Septal Ablation
  Other Names: Alcohol Septal Ablation
  Arms: Reference Group; Study Group

SUMMARY:
Patients with HOCM and severe LVOT obstruction can remain asymptomatic while significant cellular and structural changes of the heart (adverse remodeling) may occur preceding heart failure and rhythm disorders. Hence, preventing adverse remodeling through LVOT desobstruction may have significant impact on cardiac function and geometry in this particular population, as it is in symptomatic patients.

The investigators will assess functional and structural characteristics of the myocardium in asymptomatic vs. symptomatic patients with severe LVOT obstruction before and after PTSMA, using advanced imaging studies with LGE-CMR and echocardiography.

DETAILED DESCRIPTION:
The trial consists of three cohorts

1. Symptomatic HOCM patients with severe LVOT obstruction undergoing PTSMA (reference group)
2. Asymptomatic HOCM patients with severe LVOT obstruction undergoing PTSMA (study group)
3. Asymptomatic HOCM patients with severe LVOT obstruction with no intervention (observation group)

ELIGIBILITY:
Inclusion Criteria:

* Age > 40 yrs
* HOCM diagnosed by experienced cardiologists (European Society of Cardiology (ESC)-certified imaging cardiologists and/or finalized fellowship imaging)
* LVOT obstruction >30 mmHg pressure gradient in rest, or >50 mmHg during exercise by TTE and/or invasive measurement, performed experienced (imaging) cardiologists
* Symptomatic (NYHA class >2 or CCS class >2)
* Asymptomatic: free of any dyspnea/chest pain or discomfort associated with LVOT obstruction

Exclusion Criteria:

* LV wall thickness <15 mm
* Other conditions responsible for hypertrophy (e.g. hypertension, aortic valve disease)
* Moderate to severe mitral valve regurgitation
* Systolic anterior motion of the mitral valve
* Coronary artery disease requiring intervention
* Pregnancy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-01-21 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Fibrosis | 2 years
  Extracellular Volume Fraction
Global longitudinal strain (TTE) | 2 years
  Diastolic Function
Deformation (CMR) | 2 years
  Shortening Index
Haemodynamics | 2 years
  Left and Right-Sided Pressure Gradients (TTE)
4D velocity mapping | 2 years
  Blood Flow
LV Geometry | 2 years
  Volume

SECONDARY OUTCOMES:
New York Heart Association (NYHA) classification | 2 years
  Exercise tolerance

CONTACTS AND LOCATIONS:
Overall Officials: Jurrien M ten Berg, MD PhD, Principal Investigator — St. Antonius Hospital; Fatih Arslan, MD PhD, Principal Investigator — St. Antonius Hospital
Locations (1):
- St. Antonius Hospital, Nieuwegein, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arslan F, Akdim F, Ten Berg JM. Reverse remodeling after percutaneous transluminal septal myocardial ablation in severe but asymptomatic LVOT obstruction (RASTA) study: Rationale and design of transcatheter septal reduction in asymptomatic patients with severe hypertrophic obstructive cardiomyopathy. Catheter Cardiovasc Interv. 2021 Feb 15;97(3):488-492. doi: 10.1002/ccd.29178. Epub 2020 Aug 18. PMID 32808736